CLINICAL TRIAL: NCT06046664
Title: A Study Assessing the Impact of the Oncotype DX DCIS Score on Radiotherapy Decision Making in the United Kingdom
Brief Title: Oncotype DX DCIS: Impact on Radiotherapy Decision Making
Acronym: ONCOTYPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR4963
Record Dates: First submitted 2023-01-17; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCIS Test (Other)
  Interventions: Diagnostic Test: ONCOTYPE DX DCIS test

INTERVENTIONS:
Diagnostic Test: ONCOTYPE DX DCIS test — The Oncotype DX DCIS score, comprised of 12 of the 21 genes of the Oncotype DX Recurrence score, has been developed by Genomic Health Inc.
  Two clinical utility studies have now been performed in USA, assessing the value of the Oncotype DX DCIS to clinical decision making (18,19) The first study by Alvarado et al. evaluated the influence of the test in 10 centres and in 115 patients (18). The DCIS score led to a change in the treatment recommendation in 36 patients (31.3%; 26 patients had a change to no radiation and 10 patients had a change to recommend radiation). The second study similarly showed change in recommendations following the Oncotype DX DCIS test in 26.4% of cases. It is unclear what the impact of the DCIS score test would be in the UK.

SUMMARY:
Prospective single centre study of patients with DCIS that have undergone breast conservation surgery.

DETAILED DESCRIPTION:
This is a single centre (Royal Marsden Hospital - Chelsea and Sutton) non-randomised trial investigating whether the Oncotype DX DCIS score changes the radiotherapy recommendation made by clinical oncologists in patients with low to moderate risk DCIS following breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of DCIS
2. DCIS treated with breast conserving surgery

Exclusion Criteria:

1. Prior treatment for DCIS or invasive breast cancer in ipsilateral breast.
2. Patients with contra-indications to radiotherapy, including prior breast radiotherapy
3. Patients who undergo mastectomy for DCIS
4. Age < 45 years old
5. Patients with > 25mm DCIS
6. Patients with multifocal DCIS (defined as more than 1 distinct focus of DCIS with at least 50mm of intervening benign tissue)
7. Patients with invasive (including microinvasion) disease
8. Patients with positive axillary nodal disease (including isolated tumour cells)
9. Patients with close (<1mm) or positive radial margins (unless maximally surgically excised or no further DCIS on re-excision)
10. Patients recommended adjuvant endocrine therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in radiotherapy recommendation by clinician | end of trial (2 years)
  Percentage of clinical oncology recommendations regarding radiotherapy that change pre- and post- Oncotype DX DCIS.

SECONDARY OUTCOMES:
Determine whether the Oncotype DX DCIS score results in a change in patient decision for adjuvant radiotherapy. | end of trial (2 years)
  Percentage of patients who change their decision regarding radiotherapy pre- and post- Oncotype DX DCIS.
Determine whether the local recurrence risk estimated by clinical oncologists agrees with the local recurrence risk calculated by the Oncotype DX DCIS score (for all recurrences and for invasive recurrences only). | end of trial (2 years)
  Agreement between the local recurrence risk estimated by clinical oncologists and the local recurrence risk calculated by the Oncotype DX DCIS score (for all recurrences and for invasive recurrences only).
Determine change in patient decisional conflict pre and post Oncotype DX DCIS. | end of trial (2 years)
  Change in patient decisional conflict scale (DCS) scores pre and post Oncotype DX DCIS
Determine change in patient anxiety pre and post Oncotype DX DCIS. | end of trial (2 years)
  Change in state anxiety and trait anxiety scores using the State Trait Anxiety Inventory (STAI) pre and post ONCOTYPE DX DCIS test
Determine patient, tumour and clinician factors that are associated with clinicians changing their decision regarding radiotherapy. | end of trial (2 years)
  Patient, tumour and clinician factors (data collected during Visit 1) that are associated with clinicians changing their decision regarding radiotherapy.
Determine patient, tumour and clinician related factors that are associated with patients changing their decision regarding radiotherapy. | end of trial (2 years)
  Patient, tumour and clinician related factors (data collected during Visit 1) that are associated with patients changing their decision regarding radiotherapy.
Determine patient, tumour and clinician related factors that are associated with patients' final decision to have radiotherapy. | end of trial (2 years)
  Patient, tumour and clinician factors that are associated with patients' final decision to have radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No